CLINICAL TRIAL: NCT00563732
Title: An Open-Label, Nonrandomized Study to Evaluate the Potential Pharmacokinetic Interaction Between Multiple Doses of Lecozotan SR and a Single Oral Dose of Digoxin When Administered Orally to Healthy Adult Subjects
Brief Title: Study Evaluating Potential Pharmacokinetic (PK) Interaction Between Lecozotan and Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3098B1-1142
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — lecozotan

INTERVENTIONS:
Drug: Lecozotan

SUMMARY:
Primary: To evaluate the effects of multiple doses of lecozotan SR on the PK profile of a single dose of digoxin in healthy adult subjects.

Secondary: To assess the safety and tolerability of the coadministration of lecozotan SR and digoxin.

ELIGIBILITY:
Inclusion Criteria:

* Women of non childbearing potential and men aged 18 to 55 years at screening.
* Body mass index (BMI) in the range of 18 to 30 kg/m2 and body weight 50 kg (BMI = weight (kg)/[height (m)]

Exclusion Criteria:

* Presence or history of any disorder that may prevent the successful completion of the study.
* Any clinically important deviation from normal limits in physical examination, vital signs or clinical laboratory test results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effects of multiple doses of lecozotan SR on the PK profile of a single dose of digoxin in healthy adult subjects

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer